CLINICAL TRIAL: NCT05198050
Title: Letrozole Plus Misoprostol Versus Misoprostol Alone in Induction of Abortion of Anembryonic Pregnancy:
Brief Title: Letrozole in Induction of Abortion of Anembryonic Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdalla, Clinical professor of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Letrozole and abortion
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Anembryonic Pregnancy
Keywords: Letrozole; misoprostol; induction of abortion
MeSH Terms: interventions — Letrozole; Alprostadil

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single dose letrozole tablets (Active Comparator): starting from the first of January, patients will receive a single dose of letrozole (20 mg) two days, before starting misoprostol administration. Placebo tables with a similar appearance to letrozole will be administered the day before misoprostol administration and on the day of misoprostol administration.
  Interventions: Drug: Letrozole tablets; Drug: Misoprostol Tabets; Drug: Placebo tablets
- multiple dose letrozole tablets (Active Comparator): starting from the first of January, patients will receive 10 mg letrozole daily for two days before the day of misoprostol administration and on the day of misoprostol administration.
  Interventions: Drug: Letrozole tablets; Drug: Misoprostol Tabets
- misoprostol tablets (Active Comparator): starting from the first of January, patients will receive placebo tablets with a similar appearance to letrozole daily for two days before the day of misoprostol administration and on the day of misoprostol administration.
  Interventions: Drug: Misoprostol Tabets; Drug: Placebo tablets

INTERVENTIONS:
Drug: Letrozole tablets — Letrozole is a third-generation non-steroidal aromatase inhibitor
  Arms: multiple dose letrozole tablets; single dose letrozole tablets
Drug: Misoprostol Tabets — a synthetic prostaglandin medication
  Other Names: prostaglandin E1
Drug: Placebo tablets — Placebo tables with a similar appearance to letrozole
  Arms: misoprostol tablets; single dose letrozole tablets

SUMMARY:
Some studies suggest the prescription of aromatase inhibitors prior to the use of misoprostol for inducing drug abortion. the aim of the study is to compare the effectiveness of various regimens of letrozole combined with misoprostol versus using misoprostol alone in inducing complete abortion in patients with blighted ovum.

DETAILED DESCRIPTION:
Some studies suggest prescription of aromatase inhibitors prior to the use of misoprostol for inducing drug abortion, increases the efficiency of the treatment regimen and also decreases the need for surgical interventions. Some conducted studies have mentioned reinforcing the impact of misoprostol with letrozole, but reaching the ideal dose still needs more studies, so in this study, the investigators will compare the effectiveness of various regimens of letrozole ( 10 mg/d for 3 days or a single dose of 20 mg) combined with misoprostol versus using misoprostol alone in inducing complete abortion in patients with a blighted ovum.

ELIGIBILITY:
Inclusion Criteria:

* first trimester of pregnancy
* pregnancy duration less than 12 weeks based on LMP.
* non-viable fetus (blighted ovum)

Exclusion Criteria:

* No heart disease,
* No asthma
* No History of thromboembolism
* No History of cancer
* No renal failure
* No liver diseases
* History of allergy to misoprostol or letrozole drugs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Complete abortion | 2 days
  no emergency or elective curettage was necessary until next menstruation

SECONDARY OUTCOMES:
Induction-to-abortion interval | 2 days
  the interval between administration of misoprostol)
Adverse effects of Misoprostol | 2 days
  diarrhea, abdominal cramps, fever and sweating.
Adverse effects of Letrozole | 2 days
  hot flushes, drowsiness and nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Abdalla, MD, Principal Investigator — Kasralainy teaching hospital
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fouda UM, Sayed AM. Extended letrozole regimen versus clomiphene citrate for superovulation in patients with unexplained infertility undergoing intrauterine insemination: a randomized controlled trial. Reprod Biol Endocrinol. 2011 Jun 21;9:84. doi: 10.1186/1477-7827-9-84. PMID 21693030
- [Background] Abbasalizadeh F, Sahhaf F, Sadeghi-Shabestari P, Mirza-Aghazadeh-Attari M, Naghavi-Behzad M. Comparison Between Effect of Letrozole Plus Misoprostol and Misoprostol Alone in Terminating Non-Viable First Trimester Pregnancies: A Single Blind Randomized Trial. J Family Reprod Health. 2018 Mar;12(1):27-33. PMID 30647756
- [Background] Lee VCY, Ng EHY, Yeung WSB, Ho PC. Misoprostol with or without letrozole pretreatment for termination of pregnancy: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):317-323. doi: 10.1097/AOG.0b013e3182073fbf. PMID 21252745
- [Background] Lee VC, Yeung TW, Tang OS, Ng EH, Yeung WS, Ho PC. Effect of letrozole on uterine artery Doppler flow indices prior to first-trimester termination of pregnancy: a randomized controlled trial. Ultrasound Obstet Gynecol. 2012 Oct;40(4):392-7. doi: 10.1002/uog.11115. PMID 22302719